CLINICAL TRIAL: NCT05969964
Title: Can Second Resection for pT1 Bladder Carcinoma be Safely Avoided After Initial En-Bloc Resection With Negative Vertical and Horizontal Safety Margins: A Randomized Controlled Trial
Brief Title: Can Second Resection for pT1 Bladder Cancer be Avoided After Initial En-Bloc Resection With Negative Safety Margins
Status: Recruiting | Type: Observational
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Other Study IDs: MS.23.06.2435
Record Dates: First submitted 2023-07-03; First posted 2023-08-01 (Actual); Last update posted 2024-10-30 (Actual); Status verified 2024-10

CONDITIONS: Bladder Cancer Stage I
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Bladder tumor tissues resected during cystoscopy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Re_TUR: Those patients diagnosed with pT1 after initial ERBT with negative vertical and horizontal safety margins will undergo second look as endorsed by the guidelines.
  Interventions: Behavioral: Avoid second resection after initial complete resection
- No re_TUR: Those patients diagnosed with pT1 after initial ERBT with negative vertical and horizontal safety margins won't undergo second look as endorsed by the guidelines and will receive directly intravesical BCG
  Interventions: Behavioral: Avoid second resection after initial complete resection

INTERVENTIONS:
Behavioral: Avoid second resection after initial complete resection — Those patients diagnosed with pT1 after initial ERBT with negative vertical and horizontal safety margins won't undergo second look as endorsed by the guidelines.

SUMMARY:
The goal of this [ Can second resection for pT1 bladder carcinoma be safely avoided after initial En-Bloc Resection with negative vertical and horizontal safety margins ? is to assess the impact of avoiding re TUR on Recurrence free survival, progression free survival and cancer specific survival in patients with pT1 bladder cancer treated with ERBT and intravesical BCG through a RCT.

DETAILED DESCRIPTION:
Bladder cancer (BC) is the one of the most prevalent cancer in Egypt representing nearly 30% of all cancers. Approximately 75% of newly diagnosed BC present with non-muscle invasive disease (NMIBC). Initial treatment for most BCs includes transurethral resection (TUR) of the tumor to obtain tissues sufficient for histo-pathological examination to determine if the tumor reaches the muscular proprietary or not.

In the setting of non muscle invasive urothelial carcinoma (NMIBC) especially T1HG, several studies showed a benefit of performing repeat resection within 2- 6 weeks to ensure adequate resection and exclude invasion of muscle layer.

However, several issues make this recommendation ie. Re-TUR at least debatable . First, most of these recommendations are based on heterogenous studies that didn't report cancer specific survival (CSS). The risk of upstaging to muscle-invasive disease at re-TUR i did not exceed 7% in recent series . Moreover, the potential complications of re TUR that include bladder perforation and extravasation may delay administration of intravesical BCG and this delay is associated with increased risk of tumor recurrence and progression.

On the other hand, several studies have demonstrated that presence of detrusor muscle (DM) in the initial specimen is a surrogate marker of resection quality and was associated with less incidence of residual tumor at the re TUR. New techniques like En-bloc resection of bladder tumour (ERBT) entails a circumferential incision around the tumor with 5-10 mm safety margin, then proceed to deep muscle layer underneath the tumor where it is dissected using a combination of blunt dissection and laser or diathermy energy. This technique allows accurate assessment of the depth of invasion and the infiltration pattern of NMIBC and thus improving the accuracy of pathological diagnosis.

Recently published articles on this topic reported a higher rate of detrusor muscle in the specimen (96%) with enbloc compared to conventional TURB.

In a retrospective analysis of 106 patients with pT1 bladder cancer treated with ERBT, 50 patients underwent re-TUR and no significant benefits in terms of RFS and PFS to performing a reTUR in all patients with pT1 on initial ERBT.

Residual tumors were found in 6 patients (12%) and none of them were upstaged to T2 disease. Interestingly, no residual disease or recurrence overtime at the initial ERBT site in patients with negative horizontal safety margins and residual tumor was found in 2 out of 45 patients with negative vertical safety margins

Aim of Work

The aim of this study is to assess the impact of avoiding re TUR after initial enbloc resection of primary tumor with negative safety margins on recurrence free survival (RFS) ,progression free survival (PFR) and cancer specific survival (CSS ) in patients with pT1 bladder cancer through a RCT.

ELIGIBILITY:
Inclusion Criteria:

• Patients treated with ERBT and diagnosed with pT1 disease with negative vertical and horizontal safety margins at final pathology.

Exclusion Criteria:

* Large tumors not suitable for ERBT
* Residual tumor.
* Multicentric tumors ( more than 4 lesions)
* Presence of CIS.
* Positive vertical or horizontal safety margins after initial resection.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and female patients treated with ERBT and diagnosed with pT1 disease with negative vertical and horizontal safety margins at final pathology.
Sampling Method: Probability Sample
Enrollment: 370 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Impact of avoiding repeat resection on recurrence and progression free survival. | 12 month
  occurrence of new tumors or progression of the primary tumor will be compared between both groups. Tis will be assessed by both cystoscopy and MRI findings

SECONDARY OUTCOMES:
perioperative complications associated with re TURBT | 12 month
  The incidence of perioperative complications after repeat resection will be documented and compared between both groups. This outcome will be assessed using Dindo-Clavien classification.

OTHER OUTCOMES:
The financial cost associated with performing repeat resection. | 12 months
  Financial cost of repeat resection will be assessed in USD and compared between both groups.

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud Laymon, MD,MRCS, Principal Investigator — Urology &Nephrology Center, Mansoura University, Egypt
Locations (1):
- Urology and nephrology center, Mansoura University, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided